CLINICAL TRIAL: NCT00005479
Title: Measures of Postprandial Lipoproteins Are Not Associated With Coronary Artery Disease in Patients With Type 2 Diabetes Mellitus
Brief Title: Diabetes, Lipoproteins and Accelerated Vascular Disease
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CUMC ID unknown (4963); P01HL057217 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Atherosclerosis; Carotid Artery Diseases; Diabetes Mellitus, Non-insulin Dependent; Diabetes Mellitus
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Atherosclerosis; Carotid Artery Diseases; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
To better understand the excess cardiovascular disease associated with diabetes mellitus.

DETAILED DESCRIPTION:
BACKGROUND:

Diabetes mellitus is associated with a 2-4 fold increase in risk for atherosclerotic cardiovascular disease. Atherosclerotic cardiovascular disease, particularly coronary artery disease, is the leading cause of death in diabetics. The study was a subproject within a program project grant, with Henry Ginsberg as principal investigator. The program project was part of an institute-initiated study on The Etiology of Excess Cardiovascular Disease in Diabetes Mellitus. The initiative originated after discussions between NHLBI and the Juvenile Diabetes Foundation International (JDFI). The Request for Applications (RFA) was originally issued in October 1994 and resulted in the award of one grant The RFA was reissued in December 1995 and resulted in the awarding of five program project grants, the one under discussion among them.

DESIGN NARRATIVE:

The study, subproject 3 within a program project grant, was entitled Atherogenic Triglyceride Rich Lipoproteins in Diabetes. The subproject examined the atherogenicity of hypertriglyceridemia in subjects with non-insulin dependent diabetes mellitus (NIDDM). Subproject 3 tested hypotheses concerning the impact of the size and number of triglyceride-rich lipoproteins (TGRL) on risk for atherosclerotic cardiovascular disease (ASCVD) in several human populations. A case-control study of diabetics with or without coronary artery disease determined if TGRL size and number differed between the groups. In this study, Whites, Blacks and Hispanics with documented coronary artery disease or with less than 50 percent coronary stenosis by angiography were recruited. The hypothesis was tested that increased apoB in small TGRL was associated with coronary artery disease. Fasting and postprandial blood samples were obtained for measurement of TGRL apoB level, TGRL TG:apoB ratio, the amount of apoB in apoE-rich TGRL, and retinyl palmitate clearance. Allelic differences in the apoB, apoE, LPL, and apoCIII genes were examined for effects on the size and number of TGRL: specific hypotheses were tested regarding the impact of these alleles.

TGRL size and number were also compared in diabetics with and without carotid atherosclerosis in the Atherosclerosis Risk in Communities (ARIC) study, in Sioux and Pima Indian tribes that differed in ASCVD rates, and in Blacks, Whites and Hispanics with a range of insulin levels and insulin resistance in the Insulin Resistance and Atherosclerosis Study (IRAS). These studies served both to confirm findings in the case-control study and to provide the opportunity to investigate diverse populations. The collaboration with IRAS allowed determination of the effects of insulin resistance and insulin secretory capacity on TGRL size and number. Finally, experiments with cultured endothelial cells were performed to determine if small TGRL could cause endothelial dysfunction. PMI-1 and VCAM-1 were markers of TGRL effects. In the case-control study, plasma PMI and VCAM-1 were measured to examine their relationship to coronary artery disease and to TGRL size and number.

Dollars awarded were estimated based on the CRISP assignment of $173,249 dollars in FY 1996 for Subproject 3. This was approximately 25 percent of the total dollars awarded and was used to estimated committed dollars.

ELIGIBILITY:
Inclusion criteria

* Patients with type 2 diabetes mellitus (DM), defined by medical record diagnosis, fasting glucose >140 mg/dl, or the use of diabetes medications
* Had a myocardial infarction (MI) any time in the past, a coronary angiogram within the previous year, or an exercise perfusion scan (stress thallium study) within one year
* Patients with CAD group, defined by the following criteria: documented prior MI, PTCA/stent, CABG, or >75% stenosis in any vessel by coronary angiography.
* Patients without CAD group, defined as: the absence of a prior MI and <50% stenosis in all vessels by coronary angiography within the past year, or the combination of a normal exercise perfusion scan and the absence of a prior MI or any interventional cardiac procedures.

Exclusion criteria

* MI or cardiac procedures within the past 3 months
* Diagnoses of cancer, severe congestive heart failure (ejection fraction < 20%), kidney or liver disease, pancreatitis, other gastrointestinal conditions,
* Laboratory values of creatinine levels > 1.3, abnormal liver function tests, abnormal CBC, fasting TG > 400 mg/dl, urine protein > 2+ on urinalysis or > 1000 mg/24 h, abnormal thyroid function tests, body mass index (BMI) > 34 for men and > 37 for women or BMI < 20 for both sexes
* Age < 35 or > 75 years

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with type 2 diabetes mellitus (DM) with or without coronary artery disease (CAD)
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 1996-09; Primary Completion 2001-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Ginsberg, MD, Principal Investigator — Herbert and Florence Irving Professor of Medicine; Director, Irv, Dept Medicine Preventive Medicine
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- Available data/document: NCBI website — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2724776/